CLINICAL TRIAL: NCT02784041
Title: Comparison of the Effect of Single Adductor-canal-block and Peri-articular Infiltration on the Outcome After Unilateral Total Knee Arthroplasty
Brief Title: Single Adductor-canal-block Versus Peri-articular Infiltration on Outcome After Total Knee Arthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ZS-980
Record Dates: First submitted 2016-05-15; First posted 2016-05-26 (Estimated); Last update posted 2017-04-06 (Actual); Status verified 2016-04

CONDITIONS: Osteoarthritis,Knee
Keywords: knee arthroplasty; adductor canal block; periarticular infiltration
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- single adductor-canal-block (Experimental): Patients in this group will receive ultrasound guided single adductor-canal- block with 0.35% ropivacaine 25ml.
  Interventions: Drug: single adductor-canal-block
- periarticular infiltration (Experimental): patients in this group will receive periarticular infiltration of local anesthetic.
  Interventions: Drug: periarticular infiltration

INTERVENTIONS:
Drug: single adductor-canal-block — Single adductor-canal-block is performed before the surgery. A 12Hz linear ultrasound transducer is placed on the medial part of the thigh with the leg slightly externally rotated. The femoral artery was identified in short axis in the adductor canal, underneath the sartorius muscle. After skin disinfection , an 18-gauge needle (B.Braun Medical, Melsungen, Germany) is inserted in-plane from the lateral side of the transducer. The needle tip was placed underneath the sartorius muscle, just lateral to the artery and saphenous nerve, using 2-3 ml of saline to ensure correct placement. 25 ml of 0.35% ropivacaine is slowly injected with repeated aspiration.
  Arms: single adductor-canal-block
Drug: periarticular infiltration — The periarticular infiltration of multimodal agents will involve the preparation of a mixture of 100 ml solution. The mixture contains 30ml (300mg) ropivacaine, 0.5ml (5 mg) morphine, 2 ml (50 mg) flurbiprofen and 0.5 ml of 1:1000 epinephrine, and then is diluted with 0.9% normal saline to a total volume of 100ml. 50 ml of mixture will be injected into the anterior, medial and lateral soft tissues after the implantation of the joint prostheses. The remaining 50 ml of mixture will be injected into intraarticular space after the closure of articular capsule.
  Arms: periarticular infiltration

SUMMARY:
The purpose of this study is to compare the effect of single adductor-canal-block versus single femoral nerve block on the recovery after total knee arthroplasty.

DETAILED DESCRIPTION:
The aim of this study is to assess the effect of different analgesic effects on the outcome of patients undergoing total knee arthroplasty. Patients who will have primary unilateral total knee replacement between September 2016 to June 2018 at Peking Union Medical College Hospital and meet the inclusion criteria will be included. They are randomized into two groups. The total knee arthroplasty is performed by one surgeon and adductor-canal block is performed by one anesthesiologist who is not responsible for follow-up. Patients on both groups will have intravenous patient control analgesia with 1 mg morphine/bolus. One residency is responsible for the follow-up.

ELIGIBILITY:
Inclusion Criteria:

* osteoarthritis
* unilateral total knee arthroplasty
* ASA grade I - II
* normal cognitive function.

Exclusion Criteria:

* patients refuse
* BMI > 35
* diagnosis other than osteoarthritis
* allergy to the drugs used or contraindication to the intervention

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2016-09; Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
the time required for functional recovery | from the date of the surgery to the time when the patients meet the criteria of functional recovery. The earliest day on which the patient achieves the criteria of functional recovery will be recorded and the average time is 7 days after surgery.
  Patients are evaluated postoperatively to determine whether the patients have meet the criteria of functional recovery.The criteria of functional recovery are as followings: walking distance more than 70m with crutch, getting up or standing up independently and visual analog score less than 5 both in rest and after movement. Before discharge, patients are assessed every morning. After discharge, patients are followed up by phone every two days.

SECONDARY OUTCOMES:
postoperative WOMAC scales | pre-operative, three months,six months and one year afer the surgery
  We compare the WOMAC scales of two groups before, three months, six months, and one year after the surgery.
Postoperative complications | daily after the surgery until discharge from hospital, expected average up to 5 days after the surgery
  Any complication, including nause and vomiting, deep vein thrombosis, pulmonary embolism, pulmonary infection, urinary tract infection,cardiovascular event and falls are recorded during inhospital stay.
postoperative VAS scale | pre-operative, 6h postoperative, 24h postoperative, 48h postoperative, one month postoperative, three-month postoperative, one year postoperative
  Pain at rest and while moving are evaluated by a visual analog scale preoperative, 6h, 24h, 48h, 1month, 3 months and 1 year after the surgery.
postoperative morphine consumption | 6h, 24h, 48h after the surgery
  Consumptions of morphine are recorded at 6h, 24h, 48h after the surgery.
postoperative SF-36 score | pre-operative, three months,six months and one year afer the surgery
  We compare the SF-36 score of two groups before, three months,six months and one year after the surgery.

OTHER OUTCOMES:
patients' satisfaction | before discharge, usually 3-4 days after the surgery and one year after the surgery
  The degree of satisfaction with surgery outcomes is assessed on a scale from fully satisfied to dissatisfied .

CONTACTS AND LOCATIONS:
Overall Officials: Yuguang Huang, Dr, Study Chair — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes